CLINICAL TRIAL: NCT03503240
Title: Patient Satisfaction With Appearance, Scar Outcome and Quality of Life After Skin Cancer Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-168
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Skin Cancer
Keywords: Quality of Life; survey; 18-168
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate patient satisfaction and quality of life as it relates to skin cancer surgery. This research study involves taking a one-time survey online.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age at the time of surgery.
* Had a diagnosis of a cutaneous malignancy

  * Cutaneous malignancy includes, but is not limited to basal cell carcinoma, squamous cell carcinoma, and melanoma
* Able to speak and read English
* MSK Only Cross Sectional Study: Radiation therapy patients ≥ 18 years of age who have received RT for skin cancer

Exclusion Criteria:

* Unable to speak and read English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At MSK potential participants will be identified as having undergone surgery/ treatment for the treatment of a cutaneous malignancy on the face or patients will be recruited in the clinic when they present for consultation or the day of skin surgery/ treatment.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-04-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
number of patients satisfied with facial appearance | 1 year
  Satisfaction with Facial Appearance Scale, Appearance-related Psychosocial Distress Scale and Adverse Effects Checklist using the FACE-Q Skin Cancer instrument.
number of patients satisfied with scar outcome | 1year
  Appraisal of Scars Scale, Appearance-related Psychosocial Distress Scale and Adverse Effects Checklist using the FACE-Q Skin Cancer instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Brigham and Women's Hospital (Data Collection Only), Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm